CLINICAL TRIAL: NCT06289621
Title: Brief Transdiagnostic Treatment for Anxiety Disorders and PTSD in South Africa: A Hybrid-Effectiveness-Implementation Trial
Brief Title: Brief Transdiagnostic Treatment for Anxiety Disorders and Post-traumatic Stress Disorder (PTSD) in South Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Stellenbosch (Other); Fogarty International Center of the National Institute of Health (NIH); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Kristina Korte, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P000420; K01TW012180 (NIH)
Record Dates: First submitted 2024-01-25; First posted 2024-03-04 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Anxiety Disorders; Post-traumatic Stress Disorder
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a Type 1 hybrid-effectiveness implementation trial. Study participants are randomized into the brief transdiagnostic treatment for anxiety disorders and post-traumatic stress disorder (PTSD) or an enhanced standard care control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxiety Disorders and Post-traumatic Stress Disorder (PTSD) Transdiagnostic Treatment ( FSET) (Experimental): The anxiety disorders and post-traumatic stress disorder (PTSD) transdiagnostic treatment (FSET) is brief, 5-session, cognitive-behavioral intervention designed to treat symptoms associated with anxiety disorders and PTSD. The treatment is administered by lay providers (e.g., nurses) in primary care clinics in South Africa.
  Interventions: Behavioral: False Safety Behavioral Elimination Treatment (FSET)
- Enhanced Standard Care Group (Other): The enhanced standard care group is the condition. Those in the enhanced standard care control group will receive standard care plus referrals. Upon completion of the study, they will be offered the anxiety disorder and post-traumatic stress disorder treatment (FSET).
  Interventions: Behavioral: Enhanced Standard Care

INTERVENTIONS:
Behavioral: False Safety Behavioral Elimination Treatment (FSET) — 5-session transdiagnostic treatment for anxiety disorders and post-traumatic stress disorder (PTSD)
  Arms: Anxiety Disorders and Post-traumatic Stress Disorder (PTSD) Transdiagnostic Treatment ( FSET)
Behavioral: Enhanced Standard Care — Participants in the enhanced standard care control group will receive treatment as usual and a list referrals.
  Arms: Enhanced Standard Care Group

SUMMARY:
The purpose of this study is to examine the use of a brief transdiagnostic treatment for anxiety disorders and (post-traumatic stress disorder (PTSD) in South Africa. The intervention will be delivered by non-specialist providers (e.g., nurses) in primary care clinics. The brief intervention group will be compared to an enhanced standard care control group.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) and anxiety disorders are highly prevalent and a leading cause of disability in low and middle-income countries (LMICs). Despite the development of evidence-based treatments (EBTs), an overwhelming majority of those in need (i.e., 85%) in LMICs do not receive treatment and, when they do, it is not empirically based. Despite the clear need for EBTs in LMICs, there are three primary barriers associated with the implementation of EBTs in these areas. These barriers include: (1) EBTs tend to be single disorder focused only treating one disorder at a time, (2) they are long in duration (e.g., 12-16 treatment sessions to treat one disorder), and (3) they tend to be complex and require a high level of skill to administer. Given the low availability of highly trained providers in LMICs, using an approach that is brief, culturally congruent, and less complex than typical EBTs is ideal for reducing these barriers. The current study aims to evaluate the use of a brief transdiagnostic treatment for anxiety disorders and PTSD (False Safety Behavior Elimination Treatment; F-SET) in South African primary care clinics. The current study is a Type 1 hybrid effectiveness-implementation trial assessing the effectiveness of the adapted brief transdiagnostic intervention and to explore facilitators and barriers to implementation. The adapted intervention is being compared to an enhanced standard care control condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with a primary anxiety disorder (panic disorder, generalized anxiety disorder, social anxiety disorder, or obsessive-compulsive disorder) or post-traumatic stress disorder.

Exclusion Criteria:

* Participants who are acutely suicidal, have severe alcohol of substance use disorder, or are engaged in another form of psychotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Structured Clinical Interview for the DSM-5 (SCID-5) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Diagnostic assessment assessing the presence or absence of a mental health diagnosis.
Clinician-Administered PTSD Scale for the DSM-5 (CAPS) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Diagnostic assessment assessing the presence or absence of post-traumatic stress disorder (PTSD)
Work Social Adjustment Scale (WSAS) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Assessment of functional impairment. Scores range from 0 to 40 with higher scores indicating higher levels of functional impairment.
General Anxiety Disorder-7 (GAD-7) | pre-treatment, immediately after the last treatment session, and 3-month follow-up
  General measure of anxiety. Scores range from 0 to 21 with higher scores indicating greater level of anxiety.
Beck Anxiety Inventory (BAI) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Measure of anxiety symptoms. Scores range from 0 to 63 with higher scores indicating greater levels of anxiety.
Safety Aid Scale (SAS) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Assessment of safety aid utilization and avoidance in anxiety disorders and PTSD. Higher scores indicate greater safety aid utilization.

SECONDARY OUTCOMES:
Post-traumatic Disorder Checklist (PCL-5 PTSD Checklist (PCL-5) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  PTSD symptom measure. Scores range from 0 to 80 with higher scores indicating greater level of post-traumatic stress symptoms.
Patient Health Questionnaire - 9 (PHQ-9) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Measure of emotional distress. Scores range from 0 to 20 with higher scores indicating greater emotional distress.
Beck Depression Inventory (BDI) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Measure of depressive symptoms. Scores range from 0 to 63 with higher scores indicating greater levels of depression.
Anxiety Sensitivity Index -3 | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Assessment of anxiety sensitivity. Scores range from 0 to 72 with higher scores indicated higher levels of anxiety sensitivity.

OTHER OUTCOMES:
Life Events Checklist (LEC) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Assessment of exposure to traumatic events. Endorsement of events indicates the degree to which one has been exposed to traumatic events.
Alcohol Use Disorders Identification Test (AUDIT) | pre-treatment, post-treatment (immediately after the last treatment session), and 3-month follow-up
  Assessment of alcohol use. Scores range from 0 to 40 with higher scores indicating possible problematic alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- Stellenbosch University, Cape Town, South Africa

REFERENCES:
- [Background] Riccardi CJ, Korte KJ, Schmidt NB. False Safety Behavior Elimination Therapy: A randomized study of a brief individual transdiagnostic treatment for anxiety disorders. J Anxiety Disord. 2017 Mar;46:35-45. doi: 10.1016/j.janxdis.2016.06.003. Epub 2016 Jun 18. PMID 27397584
- [Background] Korte KJ, Norr AM, Schmidt NB. Targeting Safety Behaviors in the Treatment of Anxiety Disorders: A Case Study of False Safety Behavior Elimination Treatment. Am J Psychother. 2018 Jul 1;71(1):9-20. doi: 10.1176/appi.psychotherapy.20180001. Epub 2018 May 7. PMID 29733676
- [Background] Schmidt NB, Buckner JD, Pusser A, Woolaway-Bickel K, Preston JL, Norr A. Randomized controlled trial of false safety behavior elimination therapy: a unified cognitive behavioral treatment for anxiety psychopathology. Behav Ther. 2012 Sep;43(3):518-32. doi: 10.1016/j.beth.2012.02.004. Epub 2012 Mar 9. PMID 22697441